CLINICAL TRIAL: NCT01098448
Title: Control of Periodontal Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Forsyth Institute (Other)
Collaborators: Göteborg University (Other); Boston University (Other)
Responsible Party: Sigmund Socransky, The Forsyth Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NIDCR-012861
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Periodontitis
Keywords: Amoxicillin; antibiotics; chronic periodontitis; local drug delivery; metronidazol; randomized controlled trial; subgingival scaling; surgery; tetracycline; moderate to advanced chronic periodontitis
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing; Amoxicillin; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Scaling and root planing (Active Comparator): scaling and root planing as a solo therapy
  Interventions: Other: scaling and root planing
- Periodontal surgery (Experimental)
  Interventions: Other: surgery
- systemic antibiotics (Experimental)
  Interventions: Drug: systemic metronidazole and amoxicillin
- Local delivery of tetracycline (Experimental)
  Interventions: Drug: local tetracycline
- local antibiotic and systemic antibiotics (Experimental)
  Interventions: Drug: local antibiotics and systemic metronidazole and amoxicillin
- local antibiotics and surgery (Experimental)
  Interventions: Other: local tetracycline and periodontal surgery
- systemic antibiotics and surgery (Experimental)
  Interventions: Other: periodontal surgery and systemic metronidazole and amoxicillin
- local and systemic antibiotics and surgery (Experimental)
  Interventions: Other: surgery, local tetracycline, systemic metronidazole and amoxicillin

INTERVENTIONS:
Other: scaling and root planing — scaling and root planing as a single therapy
  Arms: Scaling and root planing
Drug: local tetracycline — local delivery of tetracycline fibers releasing approximately 1.7 mg/tooth in all pockets >5mm
  Arms: Local delivery of tetracycline
Drug: systemic metronidazole and amoxicillin — systemic metronidazole (250 mg tid x 14) and amoxicillin (500 mg bid x 14
  Arms: systemic antibiotics
Other: surgery — periodontal surgery in residual pockets of >4mm
  Arms: Periodontal surgery
Drug: local antibiotics and systemic metronidazole and amoxicillin — 1.7 mg/tooth tetracycline fiber plus metronidazole (250 mg tid x14d)and amoxicillin (500 mg bid x 14d)
  Arms: local antibiotic and systemic antibiotics
Other: local tetracycline and periodontal surgery — local delivery of tetracycline fibers releasing approximately 1.7 mg/tooth in all pockets >5mm and periodontal surgery in residual pockets of >4mm
  Arms: local antibiotics and surgery
Other: periodontal surgery and systemic metronidazole and amoxicillin — surgery in residual pockets >4mm and metronidazole (250mg tidx14d) and amoxicillin (500mg bidx14d)
  Arms: systemic antibiotics and surgery
Other: surgery, local tetracycline, systemic metronidazole and amoxicillin — periodontal surgery in residual pockets >4mm, tetracycline ibers releasing approximately 1.7 mg/tooth in pockets >5mm, systemic metronidazlo (250mg tidx14d) and amoxicillin (500 mg bidx14d)
  Arms: local and systemic antibiotics and surgery

SUMMARY:
The purpose of this study is to test combined effects of scaling and root planing with periodontal surgery, systemically administered amoxicillin and metronidazole, and/or local tetracycline on pocket depth reduction and attachment level "gain" in patients with chronic periodontitis.

DETAILED DESCRIPTION:
In this 2x2x2 factorial design study, 229 moderate to advanced chronic periodontitis patients stratified according to current smoking status were recruited in USA and Sweden. Patients were randomly assigned to 8 groups, all of which were treated by SRP plus none, one, two or three adjunctive treatments. Thus, patients were assigned to groups that did or did not receive Surg, LAb, SAb or LAb+SAb (All) providing 8 treatment combinations (Surg + All, Surg + SAb, Surg + LAb, Surg alone, SRP + All, SRP + SAb, SRP + LAb, SRP alone). Clinical, microbiological and immunological measurements were taken for 2 years (at baseline, 3, 6, 12, 18 and 24 months). To focus on changes diseased sites, analysis was restricted to sites with baseline pocket depth greater than 5 mm. (also, these were the only sites treated by LAb). In this report, main effects and interactions were evaluated for PD reduction and AL gain two years post therapy for 187 of patients. Mean values were computed for each treatment group and averages after 2 years were compared to baseline by ANOVA. Factorial ANCOVA was used to examine significance of differences between Surg or not, SAb or not and LAb or not for PD reduction and AL gain using baseline attachment level or pocket depth as covariates and including current smoking as a factor.

ELIGIBILITY:
Inclusion Criteria:

* greater than 20 years of age
* had a least 15 natural teeth
* in good general health
* at least 4 teeth with pockets > 6 mm
* at least 8 teeth with AL > 3 mm at baseline

Exclusion Criteria:

* pregnant or nursing (if female)
* having antibiotic or periodontal therapy in the previous three months
* systemic conditions that would affect the course of periodontal disease
* systemic conditions that required antibiotic coverage
* allergic to drugs used in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 1999-09; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level Gain | 24 months

SECONDARY OUTCOMES:
Probing pocket depth reduction | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: J Max Goodson, DDS, PhD, Principal Investigator — The Forsyth Institute; Anne D Haffajee, BDS, Principal Investigator — The Forsyth Institute
Locations (1):
- The Forsyth Institute, Boston, Massachusetts, United States